CLINICAL TRIAL: NCT03547518
Title: Sham Controlled Trial of Rapid Induction Percutaneous Tibial Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Professor and Chairman, Department of Urology, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-497
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Overactive Bladder
Keywords: Urinary Urgency; Urinary Frequency; Urge Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Intervention Model Description: Randomized, single blind parallel assignment
Who Masked: Participant
Masking Description: Participant blinded to interventional or sham treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active PTNS treatment (Experimental): One-week induction consisting of three active PTNS treatments, each 2 hours long
  Interventions: Device: PTNS treatment
- Sham treatment (Sham Comparator): One-week induction consisting of three sham treatments, each 2 hours long
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: PTNS treatment — One-week induction consisting of three active PTNS treatments, each 2 hours long
  Other Names: Urgent PC Neuromodulation System
  Arms: Active PTNS treatment
Device: Sham treatment — One-week induction consisting of three active PTNS treatments, each 2 hours long
  Other Names: Simulated treatment
  Arms: Sham treatment

SUMMARY:
The aim of this study is to determine the efficacy of an accelerated course for percutaneous tibial nerve stimulation (PTNS) induction to treat overactive bladder symptoms. The standard 12 weekly induction treatments may be a patient burden and a more rapid induction may speed up symptomatic improvement.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a common condition with a prevalence ranging from 5.9% to 16.9% in the United States and has been found to increase with age. OAB has a negative impact on health related quality of life (QoL), Per American Urological Association (AUA) / Society of Urodynamics, Female Pelvic Medicine and Urogenital Reconstruction (SUFU) guidelines, PTNS is a third line recommendation for OAB along with onabotulinumtoxinA (BTX) injection and sacral neuromodulation. In the single sham-controlled trial (SUmiT: n=220), Peters et al reported that 54.5% of PTNS subjects had moderately or markedly improved bladder symptoms on global response assessments (GRA) compared to 20.9% of sham subjects (p <0.001). PTNS subjects also had statistically significant improvements in frequency, nighttime voids, voids with moderate to severe urgency and urge urinary incontinence (UUI) episodes compared to sham. There is also early data from an implanted chronic tibial nerve stimulation lead study that shows a minimum of 8 hours of tibial nerve stimulation a day results in significant improvement in incontinence episodes per day at one week. Our study will test the concept of whether the PTNS effect is dose (total time of treatment) sensitive, and whether expanding the dosage of each treatment, i.e. from 30 minutes to 2 hours, will provide significant clinical improvement after a one week induction course.

ELIGIBILITY:
Inclusion Criteria:

* Women and men > 18 years of age
* Self-reported failed conservative care of behavioral modifications and/or oral medications
* An above normal urinary frequency as recorded on initial 3-day voiding diary
* Self-reported bladder symptoms greater than or equal to 3 months
* On a stable dose of antimuscarinics/beta-3 agonists for greater than or equal to 4 weeks, and willing to remain on the medication for the duration of the study OR discontinued antimuscarinics/beta-3 agonists for greater than or equal to 2 weeks
* Capable of giving informed consent
* Ambulatory and able to use toilet independently without difficulty
* Capable and willing to follow all study-related procedures

Exclusion Criteria:

* Pregnant or planning to become pregnant during study duration
* Diagnosis of neurogenic bladder
* Botox use in bladder or pelvic floor muscles within past 12 months
* Pacemakers or implantable defibrillators
* Current urinary tract infection
* Active use of neuromodulation in any other form. If patient has InterStim, must be turned off for 2 weeks for a washout period and remain off during the entirety of the study.
* Current use of Transcutaneous Electrical Nerve Stimulation (TENS) in pelvic region, back or legs
* Previous PTNS treatment who received greater than 6 treatments. Those who have received less than 6 treatments will be allowed to screen if the last treatment was at least 6 months prior to screening.
* Use of investigational drug/device therapy within past 4 weeks
* Participation in any clinical investigation involving or impacting gynecologic, urinary or renal function within past 4 weeks
* Current or past history of any physical condition that, in the investigator's opinion, might put the subject at risk or interfere with study results

Note: For the sake of preserving scientific integrity, one or more of the eligibility criteria have been left off the list posted while the trial is ongoing. A full list of eligibility criteria will be posted upon completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospitals, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was primarily through physician referrals from private urology clinics. Recruitment began in March 2018 and concluded in May 2022.
Period: Overall Study
Arm/Group | Active PTNS Treatment | Sham Treatment
Started | 13 | 12
Completed | 11 | 12
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active PTNS Treatment | Sham Treatment | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.77 (10.08) | 60.75 (8.01) | 62.32 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Improvement in GRA for Overall Bladder Symptoms
Description: Number of subjects reporting "Moderately" or "Markedly Improved" responses on the GRA after 3 interventions
Time Frame: One week post induction (+/- 3 days)
Population: One active treatment subject did not complete primary outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Active PTNS Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 12
Participants | 3 | 2

2. Secondary Outcome: Change From Baseline Urinary Frequency on 3 Day Voiding Diary
Description: Change in number of total voids as measured by 3-day voiding diary, between pre-induction (baseline) and post-induction (post-treatment). Positive change means reduction in urinary frequency from baseline, negative change means increase in urinary frequency from baseline.
Time Frame: Baseline and 1 week post induction (+/- 3 days)
Population: 1 active treatment subject did not complete the diary.
Measure: Mean (Standard Deviation); unit: number of voids
Arm/Group | Active PTNS Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 12
number of voids | 5 (6.21) | 1.08 (5.38)
Statistical Analysis 1: Comparison: Active PTNS Treatment vs Sham Treatment; Test type: Superiority; p = 0.111, t-test, 2 sided

3. Secondary Outcome: Change From Baseline Nocturia in 3 Day Voiding Diary
Description: Change in number of total night time urinary voids over three days as measured by 3-day voiding diary, between pre-induction (baseline) and post-induction (post-treatment). Positive change means reduction in number of night time voids. Negative change means increase in number of night time voids.
Time Frame: Baseline and one week post induction (+/- 3 days)
Population: 1 active subject did not complete the diary
Measure: Mean (Standard Deviation); unit: number of night time voids
Arm/Group | Active PTNS Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 12
number of night time voids | -0.64 (2.11) | 0.31 (4.05)
Statistical Analysis 1: Comparison: Active PTNS Treatment vs Sham Treatment; Test type: Superiority; p = 0.487, t-test, 2 sided

4. Secondary Outcome: Change From Baseline in Degree of Urgency in 3 Day Voiding Diary
Description: Change in number of urinary voids recorded as urgent over three days as measured by 3-day voiding diary, between pre-induction (baseline) and post-induction (end of treatment). Positive change means reduction in urge incontinence episodes. Negative change means increase in urge incontinence episodes.
Time Frame: Baseline and 1 week post induction (+/- 3 days)
Population: 1 active subject did not complete the diary
Measure: Mean (Standard Deviation); unit: number of voids recorded as urgent
Arm/Group | Active PTNS Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 12
number of voids recorded as urgent | 4.82 (9.42) | -4.38 (10.9)
Statistical Analysis 1: Comparison: Active PTNS Treatment vs Sham Treatment; Test type: Superiority; p = 0.0393, t-test, 2 sided

5. Secondary Outcome: Change From Baseline in Number of Urge Incontinence Episodes in 3 Day Voiding Diary
Description: Change in number of urge incontinence episodes over three days as measured by 3-day voiding diary, between pre-induction (baseline) and post-induction (post-treatment). Positive change means reduction in urge incontinence episodes. Negative change means increase in urge incontinence episodes.
Time Frame: Baseline and one week post induction (+/- 3 days)
Population: 1 active subject did not complete a diary
Measure: Mean (Standard Deviation); unit: number of urge incontinence episodes
Arm/Group | Active PTNS Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 12
number of urge incontinence episodes | 5 (5.66) | 2 (6.43)
Statistical Analysis 1: Comparison: Active PTNS Treatment vs Sham Treatment; Test type: Superiority; p = 0.242, t-test, 2 sided

6. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire-short Form Symptom Bother (OABq-SF)
Description: Change from baseline in total score on a 6 question survey of extent of how much patients were bothered by bladder symptoms, with each question rated on a 6 point likert scale with 1= Not at all and 6= a very great deal. Score range 0-100. Higher score equals worse overactive bladder symptoms. Positive change means improvement in OAB symptoms. Negative change means worsening of OAB symptoms.
Time Frame: Baseline and 1 week post induction (+/- 3 days)
Population: 1 active subject did not complete OABq at one week visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PTNS Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 12
score on a scale | 17.73 (18.41) | 18.97 (14.68)
Statistical Analysis 1: Comparison: Active PTNS Treatment vs Sham Treatment; Test type: Superiority; p = 0.855, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 12 weeks in active treatment group and sham treatment groups. Sham patients that continued to the open label active PTNS treatment phase were monitored for 12 weeks.
Description: Adverse events were collected at each visit by asking the participant if there were any changes to their medical history, hospitalizations, or new acute conditions.
Groups:
- Open Label Active PTNS Treatment: Sham participants that continued to the open label active PTNS treatment phase.
  One- week induction consisting of three active PTNS treatments, each 2 hours long.
Arm/Group | Active PTNS Treatment | Sham Treatment | Open Label Active PTNS Treatment
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/13 | 2/12 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active PTNS Treatment (N=13) | Sham Treatment (N=12) | Open Label Active PTNS Treatment (N=12)
Atypical Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Asthmatic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (UTI) (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Right lower extremity cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Right foot fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Right renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
COVID infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Right lower extremity tingling (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT03547518/Prot_SAP_000.pdf